CLINICAL TRIAL: NCT00356096
Title: A Phase IV Randomised, Double-blind, Placebo-controlled, Dose Titration Trial With 0.125-0.75 mg/Day Pramipexole (Sifrol®, Mirapexin®) Orally for 12 Weeks to Investigate the Safety and Efficacy in Out-patients With Idiopathic Restless Legs Syndrome Associated With Mood Disturbances
Brief Title: Phase IV Trial With Pramipexole to Evaluate Safety and Efficacy in Patients With RLS Associated With Mood Disturbances
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 248.604
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Restless Legs Syndrome; Depression
MeSH Terms: conditions — Restless Legs Syndrome; Depression | interventions — Pramipexole

INTERVENTIONS:
Drug: pramipexole

SUMMARY:
The primary objective of this study is to determine the efficacy of pramipexole 0.125 mg to 0.75 mg daily versus placebo on RLS symptoms and on associated mood disturbances and depressive symptoms, after 12 weeks of treatment

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent consistent with ICH-GCP and local IRB/IEC requirements obtained prior to any study procedures being performed and the ability and willingness to comply with study treatment regimen and to attend study assessments.
2. Male or female out-patients aged 18-80 years.
3. Diagnosis of idiopathic RLS according to the clinical RLS criteria of the IRLSSG [P03-03355]. All four criteria must be present to fulfil the diagnosis of RLS:

   An urge to move the legs, usually accompanied or caused by uncomfortable and unpleasant sensations in the legs. (Sometimes the urge to move is present without the uncomfortable sensations and sometimes the arms or other body parts are involved in addition to the legs) The urge to move or unpleasant sensations begin or worsen during periods of rest or inactivity such as lying or sitting The urge to move or unpleasant sensations are partially or totally relieved by movement, such as walking or stretching, at least as long as the activity continues The urge to move or unpleasant sensations are worse in the evening or night than during the day or only occur in the evening or night. (When symptoms are very severe, the worsening at night may not be noticeable but must have been previously present).
4. RLS symptoms present at least 2 to 3 days per week during the last 3 months prior to baseline (Visit 2).
5. In addition all of the following must be demonstrated at Visit 2 (baseline):

IRLS total score >15 A score of >=2 for item 10 of the IRLS rating scale

Exclusion Criteria:

1. Women of child-bearing potential who do not use an adequate method of contraception
2. Any women of child-bearing potential not having negative pregnancy test at screening
3. Breastfeeding women
4. Concomitant or previous pharmacologic therapy for RLS
5. All treatment less than 14 days before baseline or concomitant treatment with medication or dietary supplements, which could significantly influence RLS symptoms
6. Withdrawal symptoms of any medication must not be present at baseline
7. Previous pramipexole non-responders in other indications than RLS.
8. Hypersensitivity to pramipexole or any other component of the investigational product
9. Diagnosis of diabetes mellitus requiring insulin
10. Any of the following laboratory results at screening: clinically significant abnormalities at the investigatos discretion; Hb below lower limit of normal
11. Clinically significant renal disease at screening
12. Clinically significant hepatic disease at screening
13. Serum ferritin <10 ng/mL at screening.
14. History of/or malignant melanoma.
15. History of/or clinically significant vision abnormalities
16. History of/or any other sleep disorder
17. History of/or major depressive disorder or any psychotic disorder, mental disorders or any present Axis I psychiatric disorder according to DSM IV requiring any medical therapy, or BDI-II total score >28
18. History of/or clinical signs of suicidal behaviour, suicide ideation or acute suicidal tendency according to the investigators opinion
19. History of/or alcohol abuse or drug addiction within the last 2 years before screening
20. Patients on a shift-work-schedule or otherwise unable to follow a regular sleep-wake cycle
21. Participation in an investigational drug study within one month prior to the start of this study
22. Patients with any clinically significant conditions that in the opinion of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2006-07; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change from baseline after 12 weeks of treatment in: IRLS total score, IRLS item 10 score and BDI-II total score | 12 weeks

SECONDARY OUTCOMES:
The following endpoints will be analysed: CGI-I, IRLS and BDI-II responder rate, VAS score for pain in limbs, RLS-6 item scores, HADS-A score, RLS-QoL score, PGI responder rate, Adverse events profile, Systolic and diastolic blood pressure, Pulse rate | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (54):
- Finland (4):
  - 248.604.35801 Boehringer Ingelheim Investigational Site, Espoo
  - 248.604.35805 Boehringer Ingelheim Investigational Site, Helsinki
  - 248.604.35803 Boehringer Ingelheim Investigational Site, Lahti
  - 248.604.35802 Boehringer Ingelheim Investigational Site, Oulu
- France (7):
  - 248.604.3301A HOP Le Vinatier,Psychiat,Bron, Bron
  - 248.604.3304B Hôpital Roger Salengro, Lille
  - 248.604.3307A Cabinet Médical, Montbrison
  - 248.604.3303A Hôpital Gui de Chauliac, Montpellier Cédex 5
  - 248.604.3303C Hôpital Gui de Chauliac, Montpellier Cédex 5
  - 248.604.3302A Hôpital Pitié Salpétrière, Paris Cédex 13
  - 248.604.3305B Hôpital du Haut Levêque, Pessac Cédex
- Germany (11):
  - 248.604.4902 Boehringer Ingelheim Investigational Site, Berlin
  - 248.604.4904 Boehringer Ingelheim Investigational Site, Berlin
  - 248.604.4905 Boehringer Ingelheim Investigational Site, Berlin
  - 248.604.4906 Boehringer Ingelheim Investigational Site, Berlin
  - 248.604.4909 Boehringer Ingelheim Investigational Site, Chemnitz
  - 248.604.4901 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 248.604.4903 Boehringer Ingelheim Investigational Site, Hellersdorf
  - 248.604.4907 Boehringer Ingelheim Investigational Site, Kassel
  - 248.604.4910 Boehringer Ingelheim Investigational Site, Leipzig
  - 248.604.4908 Boehringer Ingelheim Investigational Site, Marburg
  - 248.604.4911 Boehringer Ingelheim Investigational Site, München
- Ireland (2):
  - 248.604.35305, Carrigtohill
  - 248.604.35302 Boehringer Ingelheim Investigational Site, Castledermot
- Italy (7):
  - 248.604.3901 Università degli Studi di Bologna, Bologna
  - 248.604.3905 Casa di Cura Villa Serena, Città S. Angelo (PE)
  - 248.604.3906 Clinica Psichiatrica, Pisa
  - 248.604.3902 IRCCS San Raffaele, Roma
  - 248.604.3909 IRCCS Fondazione "Salvatore Maugeri", Telese Terme (be)
  - 248.604.3908 Azienda Sanitaria San Giovanni Battista, Torino
  - 248.604.3904 IRCCS Oasi Maria SS, Troina (Enna)
- South Korea (4):
  - 248.604.82001 Boehringer Ingelheim Investigational Site, Daegu
  - 248.604.82003 Boehringer Ingelheim Investigational Site, Incheon
  - 248.604.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 248.604.82004 Boehringer Ingelheim Investigational Site, Seoul
- Spain (6):
  - 248.604.3401, Madrid
  - 248.604.3403, Madrid
  - 248.604.3405, Madrid
  - 248.604.3407, Oviedo
  - 248.604.3402, San Cugat Del Vallés (Barcelona)
  - 248.604.3404 Hospital de Donostia, San Sebastián
- Sweden (6):
  - 248.604.4602 Boehringer Ingelheim Investigational Site, Gothenburg
  - 248.604.4603 Boehringer Ingelheim Investigational Site, Gothenburg
  - 248.604.4601 Boehringer Ingelheim Investigational Site, Hedemora
  - 248.604.4605 Boehringer Ingelheim Investigational Site, Örebro
  - 248.604.4604 Boehringer Ingelheim Investigational Site, Skövde
  - 248.604.4606 Boehringer Ingelheim Investigational Site, Stockholm
- United Kingdom (7):
  - 248.604.44004 Boehringer Ingelheim Investigational Site, Cambridge
  - 248.604.44006 Boehringer Ingelheim Investigational Site, Chorley
  - 248.604.44001 Boehringer Ingelheim Investigational Site, London
  - 248.604.44007 Boehringer Ingelheim Investigational Site, Manchester
  - 248.604.44009 Boehringer Ingelheim Investigational Site, Reading
  - 248.604.44002 Boehringer Ingelheim Investigational Site, Romford
  - 248.604.44005 Boehringer Ingelheim Investigational Site, West Green, Crawley

REFERENCES:
- [Derived] Hornyak M, Sohr M, Busse M; 604 and 615 Study Groups. Evaluation of painful sensory symptoms in restless legs syndrome: experience from two clinical trials. Sleep Med. 2011 Feb;12(2):186-9. doi: 10.1016/j.sleep.2010.11.007. Epub 2011 Jan 21. PMID 21256799